CLINICAL TRIAL: NCT02145650
Title: Spasticity Registry Evaluating Epidemiology, Treatment Patterns and Clinical Needs
Acronym: STRETCh
Status: Withdrawn | Type: Observational
Why Stopped: Study suspended due to company decision prior to enrollment.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: EPI-SPAS-001
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Muscle Spasticity
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Participants: Patients with a diagnosis of CP, MS, Stroke, SCI, or TBI will be evaluated for spasticity by their healthcare provider. Patients diagnosed with spasticity requiring treatment will be enrolled in the study. There is no intervention administered in this study.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — There is no intervention administered in this study.

SUMMARY:
This study will examine the epidemiology (incidence and control of a disease), burden, clinical need, and treatment patterns of spasticity in patients with a diagnosis of Cerebral Palsy (CP), Multiple Sclerosis (MS), Stroke, Spinal Cord Injury (SCI), or Traumatic Brain Injury (TBI).

ELIGIBILITY:
Inclusion Criteria:

-Diagnosis of Cerebral Palsy (CP), Multiple Sclerosis (MS), Stroke, Spinal Cord Injury (SCI), or Traumatic Brain Injury (TBI) for a minimum of 3 months

Exclusion Criteria:

-Participation in a spasticity clinical trial in the past 5 years.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of CP, MS, Stroke, SCI, or TBI in clinical practice evaluated for spasticity.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Investigator Assessment of Spasticity Severity using a 5-Point Scale | Day 1
Percentage of Participants with Spasticity not Receiving Treatment | Day 1
Spasticity Symptom Assessment Score using a 21-item Questionnaire | Day 1
Spasticity Impact Assessment Score using a 32-item Questionnaire | Day 1

SECONDARY OUTCOMES:
Percentage of Participants with Spasticity Receiving Treatment | Day 1
Referral Patterns for Spasticity Management | Day 1
Spasticity Screening Tool Score using a 13-item Questionnaire | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Toms River, New Jersey, United States